CLINICAL TRIAL: NCT00149825
Title: Combining Antidepressant Medication and Psychotherapy for Insomnia to Improve Depression Outcome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Rachel Manber, Dr. Rachel Manber, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R21MH066131 (NIH); R21MH066131 (NIH); DSIR 83-ATAS
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2009-10-14 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Major Depressive Disorder; Insomnia
Keywords: Major Depressive Disorder; Insomnia; Sleep; Mental Health
MeSH Terms: conditions — Depressive Disorder, Major; Sleep Initiation and Maintenance Disorders; Psychological Well-Being | interventions — Escitalopram; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- MED+CBTI (Experimental): Escitalopram plus Cognitive Behavioral Therapy for Insomnia
  Interventions: Drug: Escitalopram; Behavioral: CBTI
- MED+CTRL (Active Comparator): Escitalopram plus Pseudo-desensitization Therapy for Insomnia
  Interventions: Drug: Escitalopram; Behavioral: CTRL

INTERVENTIONS:
Drug: Escitalopram — 5 to 20 mg for 12 weeks
  Other Names: Escitalopram plus Cognitive behavioral Therapy; Escitalopram plus Pseudo-desensitization Therapy
Behavioral: CBTI — Cognitive Behavioral Treatment for Insomnia
  Other Names: Cognitive Behavioral Treatment for Insomnia
  Arms: MED+CBTI
Behavioral: CTRL — Control Therapy consists of Pseudo-desensitization Therapy for Insomnia
  Other Names: Pseudo-desensitization Therapy for Insomnia
  Arms: MED+CTRL

SUMMARY:
This study will examine the effectiveness of a combination of antidepressant medication and sleep-focused psychotherapy to simultaneously treat sleep difficulties and depression.

DETAILED DESCRIPTION:
Difficulties falling and/or staying asleep are common in people who suffer from depression. Persistent insomnia can hinder response to treatment. In addition, individuals whose insomnia does not resolve with standard antidepressant therapy are at increased risk for recurrence of their depression. Between 60% and 84% of people who have major depressive disorder report symptoms of insomnia. This study will assess the efficacy of combining antidepressant medication and sleep-focused psychotherapy to simultaneously treat sleep difficulties and depression.

Participants in this double-blind study will be randomly assigned to receive either desensitization therapy or cognitive behavioral therapy to target insomnia. All participants will also receive escitalopram oxalate, an antidepressant medication. The study will last 12 weeks. The severity of participants' depression and insomnia will be assessed. Study visits will occur weekly for the first 6 weeks, bi-weekly for the last 6 weeks, and once 6 months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder
* HRSD(17) score of at least 14
* Presence and complaint of insomnia for at least 1 month
* Fluent in English
* Use of an effective form of contraception throughout the study

Exclusion Criteria:

* Other psychiatric disorders (e.g., bipolar disorder, post traumatic stress disorder, obsessive compulsive disorder, eating disorder)
* Psychotic symptoms
* Serious, unstable, or terminal medical condition
* Axis II diagnosis of antisocial, schizotypal, or severe borderline personality disorder
* Substance abuse
* Not willing to end other psychiatric treatment
* Previous electroconvulsive therapy or vagus nerve stimulation treatment during the last year
* Sleep apnea, restless leg, or periodic limb movement disorder (to be ruled out after first sleep study)
* Other sleep disorders
* Currently pregnant or breastfeeding
* History of seizure disorder
* Disease or condition that produces altered metabolism or hemodynamic responses
* Liver or kidney dysfunction
* Current use of any over the counter medications or herbs for mood or sleep benefits (e.g., melatonin, valerian, kava, hop extract, St. John's Wort, SAMe)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Manber, PhD, Principal Investigator — Stanford University Medical School, Department of Psychiatry and Behavioral Sciences
Locations (1):
- Stanford University, Palo Alto, California, United States

REFERENCES:
- [Background] Ong JC, Gress JL, San Pedro-Salcedo MG, Manber R. Frequency and predictors of obstructive sleep apnea among individuals with major depressive disorder and insomnia. J Psychosom Res. 2009 Aug;67(2):135-41. doi: 10.1016/j.jpsychores.2009.03.011. Epub 2009 Apr 25. PMID 19616140
- [Result] Manber R, Edinger JD, Gress JL, San Pedro-Salcedo MG, Kuo TF, Kalista T. Cognitive behavioral therapy for insomnia enhances depression outcome in patients with comorbid major depressive disorder and insomnia. Sleep. 2008 Apr;31(4):489-95. doi: 10.1093/sleep/31.4.489. PMID 18457236

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between June 2004 and August 2006 through newspaper advertisements, electronic bulletin boards, community postings, and brochures in clinics.
Pre-assignment Details: Enrolled participants were screened to determine if inclusion exclusion criteria were met. This process included structured clinical interviews, completion of sleep logs, and an ambulatory screening sleep study to rule out other sleep disorders.
Groups:
- MED+CTRL: Escitalopram plus control therapy for insomnia in depression
Period: Overall Study
Arm/Group | MED+CBTI | MED+CTRL
Started | 15 | 15
Completed | 10 | 12
Not Completed | 5 | 3
Not completed — Intolerance to medication side effects | 1 | 2
Not completed — Time commitments | 2 | 1
Not completed — Not liking insomnia therapy | 1 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MED+CBTI | MED+CTRL | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 27
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (13.6) | 47.8 (13.4) | 48.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Remission of Depression (%)
Description: Percent of participants in depressive remission at 12 weeks. Remission of depression was required both an HRSD score ≤ 7 and absence of the two core symptoms of MDD based on the depression module of the SCID.
  The HRSD (Hamilton Rating of Depression Scale) measure depressive symptom severity. TIt has 17 items. The score ranges between 0 and 48. A score below 7 represents minimal symptoms.
  The SCID rates 9 symptoms of depression as present or absent. The two core symptoms of depression are sadness and anhedonia (low motivation and/or enjoyment in significant life domains).
Time Frame: After 12 weeks or at the last available time point
Measure: Number; unit: percent of participants
Arm/Group | MED+CBTI | MED+CTRL
Number analyzed (Participants) | 13 | 15
percent of participants | 61.5 | 33.3
Statistical Analysis 1: Comparison: MED+CBTI vs MED+CTRL; We hypothesized that compared with MED+CTRL, a greater percent of participants randomized to MED+CBTI will experience remission of depression; Test type: Superiority or Other; p = .13, Chi-squared; This is a one-tailed test

2. Secondary Outcome: Remission of Insomnia
Description: Percent of participants in insomnia remission. Remission of insomnia was defined by an Insomnia Severity Index (ISI)score < 8. The ISI (Insomnia Severity index) scores range between 0 and 38. A score < 8 indicates absence of insomnia.
Time Frame: After 12 weeks or at the last available time point
Population: Included in the analysis were all participants who attended at least one post randomization visit.
Measure: Number; unit: percent
Arm/Group | MED+CBTI | MED+CTRL
Number analyzed (Participants) | 13 | 15
percent | 50.0 | 7.7
Statistical Analysis 1: Comparison: MED+CBTI vs MED+CTRL; We hypothesized that compared with MED+CTRL, a greater percent of participants in MED+CBTI will experience remission of insomnia; Test type: Superiority or Other; p = .05, Chi-squared

ADVERSE EVENTS:
Arm/Group | MED+CBTI | MED+CTRL
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/13 | 0/15

LIMITATIONS AND CAVEATS:
Limitations of the current pilot study include a small sample size, relative racial homogeneity, and exclusion of patients with comorbidity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No